CLINICAL TRIAL: NCT03839641
Title: Novel Approach to Assess Metabolic Flexibility in a Respiratory Chamber
Acronym: METFLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, David McDougal, Assistant Professor-Research, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PBRC 2018-029
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fat Meal First (Experimental): Arm 1 participants randomized to receive high fat meal first, and low fat meal second
  Interventions: Other: High fat meal; Other: Low fat meal
- High Fat Meal Second (Experimental): Arm 2 participants randomized to receive low fat meal first, and high fat meal second
  Interventions: Other: High fat meal; Other: Low fat meal

INTERVENTIONS:
Other: High fat meal — 60% fat meal
Other: Low fat meal — 20% fat meal

SUMMARY:
The overarching aim of this study: To determine the effect of different meal compositions (high- vs. low-fat) on metabolic flexibility as it relates to meal-stimulated change in respiratory quotient (ΔRQ1) and sleep (ΔRQ2) metabolic flexibility, as well as the time course changes in respiratory quotient, RQ (i.e., peak RQ, time to peak RQ, nadir RQ, time to nadir, slope).

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria include:

  * Healthy male or female
  * Ages 18-40 y
  * BMI between 20 kg/m2 and 30 kg/m2 (±0.5 kg/m2 will be accepted)
  * Are willing to consume pre-prepared meals
  * Are willing to maintain current physical activity, sleep schedule, and dietary habits during the study.
  * Medically cleared for participation in the study by Medical Investigator

Exclusion Criteria:

* Participants are ineligible to participate (or will be excluded from participating in this study) if they meet any of the following criteria:

  * Unstable weight in the last 3 months [gain or loss >7 lb (or 3.2 kg)]
  * Currently working shift work
  * Smoking or use of tobacco products within the last 3 months
  * Amenorrhea (or absence of regular monthly cycles)
  * History of clinically diagnosed diabetes or a fasting blood glucose >126 mg/dL
  * Average screening blood pressure >140/90 mmHg
  * Previous bariatric surgery (or other surgeries) for obesity or weight loss
  * Use of medications affecting metabolism or sleep
  * History of neurological disease
  * History of cardiovascular disease (or other chronic diseases)
  * Pregnant, planning to become pregnant, or breastfeeding
  * Adherence to special restrained diets (e.g., low-carbohydrate, low-fat, or vegetarian/vegan diets) over the last 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- High-fat Meal, Washout (5-7 Days), and Low-fat Meal: Arm 1 participants randomized to receive high fat meal first, and low fat meal second
  High fat meal: 60% fat meal
  Low fat meal: 20% fat meal
- Low-fat Meal, Washout (5-7 Days), and High-fat Meal: Arm 2 participants randomized to receive low fat meal first, and high fat meal second
  High fat meal: 60% fat meal
  Low fat meal: 20% fat meal
Period: Overall Study
Arm/Group | High-fat Meal, Washout (5-7 Days), and Low-fat Meal | Low-fat Meal, Washout (5-7 Days), and High-fat Meal
Started | 5 | 5
Completed | 4 | 4
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-fat Meal, Washout (5-7 Days), and Low-fat Meal | Low-fat Meal, Washout (5-7 Days), and High-fat Meal | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7.5) | 27 (5.7) | 28 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8
baseline respiratory exchange ratio [Mean (Standard Deviation); unit: ratio] — The respiratory exchange ratio refers to the proportion of macronutrients being oxidized. A respiratory exchange ratio value of 1.0 indicates only carbohydrates are being oxidized, while a ratio value of 0.7 indicates only fats are being oxidized. Intermediate values, such as 0.85, indicates that both carbohydrate and fats are being oxidized.
  ratio | 0.845 (0.018) | 0.856 (0.026) | 0.851 (0.023)

OUTCOME MEASURES:

1. Primary Outcome: Overnight Respiratory Exchange Ratio
Description: 12-h mean of respiratory exchange ratio following each meal type.
  measurement interval = 12h following start of meal (7pm)
  The respiratory exchange ratio refers to the proportion of macronutrients being oxidized. A respiratory exchange ratio value of 1.0 indicates only carbohydrates are being oxidized, while a ratio value of 0.7 indicates only fats are being oxidized. Intermediate values, such as 0.85, indicates that both carbohydrate and fats are being oxidized.
Time Frame: 12 hours
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- High Fat Meal: overnight respiratory exchange ratio following high-fat meal
- Low-fat Meal: overnight respiratory exchange ratio following low-fat meal
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
ratio | 0.832 (0.014) | 0.887 (0.017)

2. Secondary Outcome: Sleep Respiratory Exchange Ratio
Description: mean of respiratory exchange ratio following each meal type during sleep period, 2am-5am., 2am-5am.
  measurement interval = 3h (2am-5am)
  The respiratory exchange ratio refers to the proportion of macronutrients being oxidized. A respiratory exchange ratio value of 1.0 indicates only carbohydrates are being oxidized, while a ratio value of 0.7 indicates only fats are being oxidized. Intermediate values, such as 0.85, indicates that both carbohydrate and fats are being oxidized.
Time Frame: 3 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
ratio | 0.820 (0.016) | 0.867 (0.034)

3. Secondary Outcome: Peak Increase in Respiratory Exchange Ratio
Description: mean of peak increase in respiratory exchange ratio (Peak values - baseline values) following each meal type
  Peak values were defined as the peak respiratory exchange ratio value measured during the post-meal period, 6pm-10pm.
  Baseline values were measured 1h prior to meal (5:00-5:45pm)
  measurement interval of peak values= 4h (6pm-10pm)
  A larger value in this measurement indicates that more carbohydrate than fats were being oxidized as fuel during the measurement period.
Time Frame: 4 h
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- High Fat Meal: change in respiratory exchange ratio following high-fat meal
- Low-fat Meal: change in respiratory exchange ratio following low-fat meal
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
ratio | 0.057 (0.030) | 0.103 (0.025)

4. Secondary Outcome: Peak Decrease in Respiratory Exchange Ratio
Description: mean of peak decrease in respiratory exchange ratio (baseline values -nadir values) following each meal type
  Peak values were defined as the peak respiratory exchange ratio value measured during the post-meal period, 6pm-10pm.
  Baseline values were measured 1h prior to meal (5:00-5:45pm)
  measurement interval of nadir values= 12h (6pm-6am)
  A larger value in this measurement indicates that more fats than carbohydrate were being oxidized as fuel during the measurement period.
Time Frame: 12 h
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
ratio | 0.093 (0.031) | 0.025 (0.038)

5. Secondary Outcome: Time to Peak Respiratory Exchange Ratio
Description: Average time from meal to peak respiratory exchange ratio value
  This measurement indicates how long on average it took form the onset of the meal, 6pm, for the participants to achieve their highest/peak respiratory exchange ratio value.
Time Frame: 12 h
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
minutes | 61.9 (13.3) | 100.3 (45.4)

6. Secondary Outcome: Time to Nadir Respiratory Exchange Ratio
Description: Average time from meal to nadir respiratory exchange ratio value
  This measurement indicates how long on average it took form the onset of the meal, 6pm, for the participants to achieve their lowest/nadir respiratory exchange ratio value.
Time Frame: 12 h
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
minutes | 274 (12.8) | 427 (113)

7. Secondary Outcome: Slope of Respiratory Exchange Ratio
Description: This value indicates the speed and magnitude of the participants change in respiratory exchange ratio between the peak and nadir values.
  A more negative value in this measurement indicates either a short time interval between the highest and lowest respiratory exchange ratio values measured and/or a large difference between the highest and lowest values of respiratory exchange ratio values measured.
Time Frame: 12 h
Measure: Mean (Standard Deviation); unit: ratio/minute
Arm/Group | High Fat Meal | Low-fat Meal
Number analyzed (Participants) | 8 | 8
ratio/minute | -0.042 (0.007) | -0.028 (0.016)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, an average of 20 days
Groups:
- High-fat Meal: High fat meal: 60% fat meal
- Low-fat Meal: Low fat meal: 20% fat meal
Arm/Group | High-fat Meal | Low-fat Meal
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-fat Meal (N=8) | Low-fat Meal (N=8)
muscle ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 1 (1)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT03839641/Prot_SAP_001.pdf